CLINICAL TRIAL: NCT00968565
Title: Regional Citrate Anticoagulation in ECMO
Brief Title: Study Using Citrate to Replace Heparin in Babies Requiring Extracorporeal Membrane Oxygenation (ECMO)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John B. Pietsch, Associate Professor of Pediatric Surgery and Pediatrics, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 090717
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2010-06

CONDITIONS: Heart Defects, Congenital; Respiratory Insufficiency
Keywords: Heart Defects, Congenital; Extracorporeal Membrane Oxygenation; Citric Acid; Heparin; Respiratory Insufficiency
MeSH Terms: conditions — Heart Defects, Congenital; Respiratory Insufficiency | interventions — Sodium Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Citrate (Experimental): Sodium citrate will be infused as the blood enters the ECMO circuit and calcium chloride will be infused as the blood leaves the ECMO circuit and enters the patient
  Interventions: Drug: sodium citrate

INTERVENTIONS:
Drug: sodium citrate — Continuous infusion of 4% sodium citrate at 300 ml/hour into ECMO circuit

SUMMARY:
The purpose of this study is to determine the safety and efficacy of citrate to provide anticoagulation of an ECMO circuit without patient anticoagulation. The standard method of providing ECMO circuit anticoagulation is the use of heparin which also anticoagulates the patient and increases the risk of patient bleeding.

DETAILED DESCRIPTION:
Extracorporeal membrane oxygenation (ECMO) is a form of extended heart/lung bypass support that has been used to treat more than 650 patients over 20 years at Vanderbilt. Over 29,000 patients have been treated worldwide. Bleeding is the most common complication during ECMO because of systemic anticoagulation with heparin. It is most commonly seen in patients following surgery either preceding or while on ECMO support. Regional citrate anticoagulation for hemodialysis was first introduced in 1961. It is the ideal alternative to heparin in patients who are at increased risk for bleeding. It permits effective anticoagulation across the extracorporeal circuit without impacting the patient's systemic coagulation. Citrate functions by binding free calcium, thereby inhibiting coagulation in both the intrinsic and extrinsic coagulation pathways. The purpose of this study is to evaluate the use of citrate as a regional anticoagulant in the ECMO circuit in high risk infants less than one year of age.

ELIGIBILITY:
Inclusion Criteria:

* Infant less than one year of age and less than 6 kg
* Informed consent obtained from parent
* One or more of the following diagnoses:
* Post-op congenital heart surgery
* Congenital diaphragmatic hernia
* Sepsis with coagulopathy not corrected prior to ECMO
* Other newborn diagnosis with Grade I or II IVH
* Infant requires/is on ECMO

Exclusion Criteria:

* Consent denied or unobtainable
* Age greater than one year
* Weight greater than 6 kg
* Gestational age less than 34 weeks

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2010-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
anticoagulation of ECMO circuit while maintaining normal coagulation and calcium levels in patient | hourly

SECONDARY OUTCOMES:
Maintain normal serum calcium levels in patients | hourly

CONTACTS AND LOCATIONS:
Overall Officials: John B Pietsch, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Background] Pinnick RV, Wiegmann TB, Diederich DA. Regional citrate anticoagulation for hemodialysis in the patient at high risk for bleeding. N Engl J Med. 1983 Feb 3;308(5):258-61. doi: 10.1056/NEJM198302033080506. No abstract available. PMID 6848936
- [Background] Bagshaw SM, Laupland KB, Boiteau PJ, Godinez-Luna T. Is regional citrate superior to systemic heparin anticoagulation for continuous renal replacement therapy? A prospective observational study in an adult regional critical care system. J Crit Care. 2005 Jun;20(2):155-61. doi: 10.1016/j.jcrc.2005.01.001. PMID 16139156
- [Background] Suzuki Y, Yamauchi S, Daitoku K, Fukui K, Fukuda I. Extracorporeal membrane oxygenation circulatory support after congenital cardiac surgery. ASAIO J. 2009 Jan-Feb;55(1):53-7. doi: 10.1097/MAT.0b013e31818f0056. PMID 19092671
- [Background] Clark JA, Schulman G, Golper TA. Safety and efficacy of regional citrate anticoagulation during 8-hour sustained low-efficiency dialysis. Clin J Am Soc Nephrol. 2008 May;3(3):736-42. doi: 10.2215/CJN.03460807. Epub 2008 Feb 13. PMID 18272829